CLINICAL TRIAL: NCT05215886
Title: Cognitive Impairment, Obesity, and the Effects of Bariatric Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1812245
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
Keywords: Obesity; Bariatric Surgery; Cognitive Screening
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery: Patients scheduled for or have already completed Weight Loss Surgery at UC Davis Medical Center
  Interventions: Behavioral: Surgery

INTERVENTIONS:
Behavioral: Surgery — Study subjects scheduled for or have already completed weight loss surgery and have already completed psychological screening as part of their pre-surgery work up

SUMMARY:
Study is designed to screen psychological cognitive baseline and retention/improvement after weight loss surgery.

DETAILED DESCRIPTION:
Patients with morbid obesity have shown to be at increased risk for memory loss and cognitive decline. Obesity and high-fat diets have been associated with deficits in learning, memory, and executive functioning. Bariatric surgery results in significant weight loss for patients and helps resolve obesity-related comorbidities such as diabetes and high blood pressure. Interestingly, bariatric surgery has shown promise in improving some aspects of cognitive function and improved memory. (3-1) Obesity affects brain structure, more specifically the grey and white matter, likely in part by reducing oxygen flow to the various regions in the brain. Studies have shown a correlation between BMI and cerebral blood flow velocity (CBFV), where higher BMI is associated with lower CBFV. Although it is not clear how exactly obesity plays a role in the brain's structural and functional changes, observations revealed compromised grey and white matter integrity, its fiber connectivity or cortical atrophy and metabolic alterations. (2)

Few studies exist on the impact of bariatric surgery on cognition. Some studies have shown that patients with obesity who underwent bariatric surgery had memory and cognitive improvement compared to those who had not undergone surgery. (4) Thus, the investigators hope to add to our understanding of how bariatric surgery can improve cognitive decline and to potentially offer surgery to more patients with baseline cognitive impairment and to improve cognitive function overall for patients with obesity. More longitudinal studies need to be done to connect bariatric surgery effects with cognitive decline, specifically memory.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive impairment/decline, memory impairment/loss, or Alzheimer's disease or dementia and bariatric surgery • Cognitive impairment/decline, memory impairment/loss, or Alzheimer's disease or dementia and obesity, and no bariatric surgery history

Exclusion Criteria:

* Patients without a history of memory impairment/loss, bariatric surgery, or obesity

  * Patients outside of University of California Davis Health System
  * Patients unable to provide consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects seeking weight loss surgery or with a history of weight loss surgery at University of California Davis Medical Center 18 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 9500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
California Verbal Learning Test-3rd Edition (CVLT-3) | Pre-operatively
  Measures episodic verbal learning including Verbal Learning, immediate memory, and delayed memory
California Verbal Learning Test-3rd Edition (CVLT-3) | 12 Months after index screening/date of surgery
  Measures episodic verbal learning including Verbal Learning, immediate memory, and delayed memory

SECONDARY OUTCOMES:
Brief Visuospatial Memory Test | Pre-operatively and 12 months after index screening/date of surgery
  Measures visuospatial learning and memory, including visual learning, immediate memory, and delayed memory.
Brief Visuospatial Memory Test | Pre-operatively
  Measures visuospatial learning and memory, including visual learning, immediate memory, and delayed memory.
Trial Making Test, A & B | 12 months after index screening/date of surgery
  Measures visual spatial attention, motor speed and cognitive flexibility
WAIS-IV Digit Span Forward & Backward | Pre-Operatively
  Measures auditory Attention (Forward), and Auditory attention and working memory (Backward)
WAIS-IV Digit Span Forward & Backward | 12 months after Index screening/date of surgery
  Measures auditory Attention (Forward), and Auditory attention and working memory (Backward)
Verbal Fluency, Phonemic & Semantic | Pre-operatively
  Measures verbal fluency by a word generation task based on letter & category (executive functioning)
Verbal Fluency, Phonemic & Semantic | 12 months after index screening/date of surgery
  Measures verbal fluency by a word generation task based on letter & category (executive functioning)
Stroop Color and Word Test; Word, Color & Word-Color | Pre-Operatively
  Measures reading speed (word), naming speed (processing) and selective attention and inhibition (attention/executive functioning)
Stroop Color and Word Test; Word, Color & Word-Color | 12 months after index screening/date of surgery
  Measures reading speed (word), naming speed (processing) and selective attention and inhibition (attention/executive functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Lyo, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan in place (yet) for data sharing

REFERENCES:
- [Result] Alosco ML, Spitznagel MB, Strain G, Devlin M, Cohen R, Paul R, Crosby RD, Mitchell JE, Gunstad J. Improved memory function two years after bariatric surgery. Obesity (Silver Spring). 2014 Jan;22(1):32-8. doi: 10.1002/oby.20494. Epub 2013 Oct 15. PMID 23625587
- [Result] Nota MHC, Vreeken D, Wiesmann M, Aarts EO, Hazebroek EJ, Kiliaan AJ. Obesity affects brain structure and function- rescue by bariatric surgery? Neurosci Biobehav Rev. 2020 Jan;108:646-657. doi: 10.1016/j.neubiorev.2019.11.025. Epub 2019 Nov 30. PMID 31794778
- [Result] Miller AA, Spencer SJ. Obesity and neuroinflammation: a pathway to cognitive impairment. Brain Behav Immun. 2014 Nov;42:10-21. doi: 10.1016/j.bbi.2014.04.001. Epub 2014 Apr 12. PMID 24727365
- [Result] Stanek KM, Gunstad J. Can bariatric surgery reduce risk of Alzheimer's disease? Prog Neuropsychopharmacol Biol Psychiatry. 2013 Dec 2;47:135-9. doi: 10.1016/j.pnpbp.2012.06.021. Epub 2012 Jul 4. PMID 22771689